CLINICAL TRIAL: NCT02885441
Title: Treatment of Acute Pancreatitis With Ketorolac
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Ilam University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Associated Professor, Ilam University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22/52/1663
Record Dates: First submitted 2016-08-23; First posted 2016-08-31 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-01

CONDITIONS: Acute Pancreatitis
Keywords: Inflammation
MeSH Terms: conditions — Pancreatitis; Inflammation | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketorolac (Experimental): Ketorolac,10 mg, 3 times daily from time of enrollment until 72 hours from enrollment for up to a maximum of 9 doses, along with the standard medical treatment
  Interventions: Drug: Ketorolac
- Control (No Intervention): The standard medical treatment

INTERVENTIONS:
Drug: Ketorolac — Ketorolac, 10 mg, 3 times daily from time of enrollment until 72 hours from enrollment. For up to a maximum of 9 doses.
  Other Names: Toradol
  Arms: Ketorolac

SUMMARY:
Patients with acute pancreatitis will be randomly assigned in either study group to receive oral (injection) Ketorolac or the control group. In patients who cannot tolerate oral medications, ketorolac injection will be used.

DETAILED DESCRIPTION:
Patients with acute pancreatitis will be randomly assigned in either study group or control group.

* The study group will receive injection or oral Ketorolac.
* The control group will receive standard medical treatment.

Ketorolac is administrated three times daily by mouth or injection starting from the time of admission for the first three days of hospitalization (72 hours).

Hs-CRP will be measured in admission in addition to standard laboratory tests.It will be done every day for up to 5 days, after the administration of study drug or till the time of discharge whichever occurs earlier. Patients will follow up for organ failure involvement and duration of hospitalization. The study will continue to gather clinical follow up information up to four months.

ELIGIBILITY:
Inclusion Criteria:

1. Predicted Severe Acute Pancreatitis
2. Enrollment within 72 hours of diagnosis
3. Obtaining informed consent
4. Age >18 years

Exclusion Criteria:

1. Heart disease, Hypertension
2. Hemorrhagic diathesis, Incomplete hemostasis, High risk of bleeding
3. Lactating women
4. Pregnancy
5. Advanced renal disease
6. Hypersensitivity to ketorolac, aspirin, other NSAIDs
7. Concurrent use with aspirin, other NSAIDs, probenecid, or pentoxifylline
8. Active or history of peptic ulcer disease
9. Recent or history of GI bleeding or perforation
10. Inflammatory bowel disease
11. Severe hepatic impairment or active hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in C-Reactive Protein (CRP) | baseline to Day 5
  baseline to Day 5

SECONDARY OUTCOMES:
Number Of Subjects With New Onset Organ Failure During Hospitalization | 30 days or until dismissal date whichever occurs earlier
  30 days or until dismissal date whichever occurs earlier
Number Of Subjects With New Onset Pancreatic Necrosis During Hospitalization | 30 days or until dismissal date whichever occurs earlier
  30 days or until dismissal date whichever occurs earlier
Duration of hospitalization | 30 days or until dismissal date whichever occurs earlier
  30 days or until dismissal date whichever occurs earlier
Mortality | 30 days or until dismissal date whichever occurs earlier
  30 days or until dismissal date whichever occurs earlier
Time of beginning and tolerance to nutrition | 30 days or until dismissal date whichever occurs earlier
  30 days or until dismissal date whichever occurs earlier

CONTACTS AND LOCATIONS:
Overall Officials: Shaahin Shahbazi, MD, Study Chair — Head of Faculty of Medicine
Locations (1):
- Ilam University of Medical Scienvc, Īlām, Iran

IPD SHARING:
Plan to Share IPD: No